CLINICAL TRIAL: NCT04822883
Title: A Single-arm, Single-blind, Multiple Dose Study to Evaluate Safety and the Effects of RL-007 on Electroencephalograms and Event-related Potentials in Subjects With Schizophrenia
Brief Title: Safety, Biomarker Study of RL-007 in Subjects With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recognify Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: C07-03-01
Record Dates: First submitted 2021-03-12; First posted 2021-03-30 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Impairment; Schizophrenia
MeSH Terms: conditions — Cognitive Dysfunction; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Four dose cohorts will be enrolled sequentially.
Who Masked: Participant
Masking Description: Participants will not be informed of their dose cohort or of the sequence of placebo or active capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose-escalation - RL-007 (Experimental): Each cohort will include a single dose-strength. Within each cohort, the sequence of active capsules and matching placebo capsules will be varied and unknown to the participant.
  Interventions: Drug: RL-007
- Dose-escalation - matching Placebo (Placebo Comparator): Within each cohort, the sequence of active capsules and matching placebo capsules will be varied and unknown to the participant.
  Interventions: Drug: RL-007 Matching Placebo

INTERVENTIONS:
Drug: RL-007 — Cohorts are 10 mg, 20 mg, 40 mg, and 80 mg with TID dosing
  Arms: Dose-escalation - RL-007
Drug: RL-007 Matching Placebo — Cohorts are 10 mg, 20 mg, 40 mg, and 80 mg with TID dosing
  Arms: Dose-escalation - matching Placebo

SUMMARY:
The purpose of this study is to assess the safety and effects on electrical activity in the brain of an investigational drug (RL-007) for improving cognition in patients with schizophrenia

DETAILED DESCRIPTION:
Potential participants will first be given an Informed Consent document and have the study explained to them. All patients who provide written informed consent will undergo screening to determine eligibility for the study. Patients who meet all eligibility criteria will be admitted to the clinic for 5 days / 4 nights as an in-patient. During this time, participants will be assigned to a specific dose cohort and will receive sequence that includes both placebo and RL-007. Brain activity and cognitive performance will be assessed on study days 2 and 4.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide a written informed consent
* Diagnosis of schizophrenia, as defined by DSM-5 and evaluated with the MINI Plus interview
* Positive and Negative Symptoms Severity Score (PANSS) of 40 - 80 (inclusive), and a score of 4 or less on the following PANSS items: P2, P3, P5, P6, G6.
* Currently being treated with a single protocol-allowed antipsychotic at a stable dose and clinically stable for at least 8 weeks before admission (note: allowed meds = aripiprazole, brexipiprazole, paliperidone, risperidone)
* Modified Simpson-Angus Scale total score <= 4
* At least 1 standard deviation below normative value of total number of words recalled on the Hopkins Verbal Learning Test
* BMI <= 38

Key Exclusion Criteria:

* History of hospitalization for medical indication within 4 weeks prior to screening or psychiatric hospitalization within 3 months prior to screening
* Use of any other psychoactive medication known to interfere with the EEG/ERP assessments within 1 week prior to screening or during the study period.
* Subjects who present a serious risk of suicide
* Any history of GI surgery, or other condition, that may affect GI absorption or any history of GI bleeding or peptic ulcer.
* Evidence or history of significant cognitive impairment, other than associated with schizophrenia, that in the judgement of the Investigator would confound secondary or exploratory assessments or prevent safe and satisfactory completion of the study protocol.
* Moderate to severe alcohol use disorder, per DSM-5 within 3 months of admission visit.
* Positive alcohol breath test or urine test for drugs of abuse at either screening or admission visit.
* Currently smoking more than 1 pack of cigarettes a day and unable or unwilling to maintain smoking to less than 1 pack a day during in-patient portion of study.
* Positive test result for SARS-CoV2 prior to admission per site standards.
* Positive test for hepatitis B, hepatitis C or HIV
* Subjects whose hair type or style is likely to interfere with successful application of scalp electrodes.
* Subjects with needle phobia or in whom venous access is technically difficult.
* Other unspecified reasons that, in the opinion of the PI or sponsor, make the subject unsuitable for enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAE) | Study Day 8.
  Comparison of AE rates between active and placebo dosing
Change in blood pressure (systolic and diastolic) from baseline | Study Day 4
  blood pressure measured in mmHg; baseline = Day -1
Change in heart rate from baseline | Study Day 4
  heart rate measured in beats per minute; baseline = Day -1
Change in respiratory rate from baseline | Study Day 4
  respiratory rate measured in breaths per minute; baseline = Day -1
Change in temperature from baseline | Study Day 4
  temperature measured in degrees Celsius; baseline = Day -1
Change in electrocardiogram (ECG) from baseline | Study Day 3
  overall physician interpretation of ECG reading; baseline = Day -1
Change in the Columbia Suicide Severity Rating Scale (C-SSRS) from baseline | Study Day 8
  The C-SSRS assesses suicidal ideation and behavior; baseline = Day -1

SECONDARY OUTCOMES:
Change from baseline in quantitative electroencephalogram (qEEG) | Study Day 4
  change from baseline in amplitude across qEEG frequency bands (alpha, beta, delta, theta, and gamma)
Change from baseline in evoked response potential (ERP) amplitude | Study Day 4
  Change from baseline in signal amplitude of the two-stimulus auditory oddball ERP
Change from baseline in evoked response potential (ERP) latency | Study Day 4
  Change from baseline in signal latency of the two-stimulus auditory oddball ERP
Change from baseline in amplitude of mismatch negativity (MMN) ERP | Study Day 4
  Change from baseline in signal amplitude of the MMN ERP
Change from baseline in latency of mismatch negativity (MMN) ERP | Study Day 4
  Change from baseline in signal latency of the MMN ERP

OTHER OUTCOMES:
Verbal learning performance | Study Day 4
  Number of words recalled (immediate and delayed) on the Hopkins Verbal Learning Test (HVLT-R)
Symbol coding performance | Study Day 4
  Number of correct responses on the Brief Assessment of Cognition in Schizophrenia Symbol Coding Test
Category fluency performance | Study Day 4
  Number of appropriate items provided in the Category Fluency Task

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, PhD, Principal Investigator — Collaborative Neuroscience Research
Locations (1):
- Collaborative Neuroscience Research, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No